CLINICAL TRIAL: NCT00326144
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo-Controlled Phase III Study of the Efficacy and Safety of Quetiapine Fumarate Sustained Release (Seroquel SR®) as Mono-Therapy in the Treatment of Adult Patients With Major Depressive Disorder
Brief Title: Efficacy and Safety of Quetiapine Fumarate Sustained Release (SEROQUEL SR) in the Treatment of Major Depressive Disorders
Acronym: OPAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1448C00003; OPAL
Record Dates: First submitted 2006-05-15; First posted 2006-05-16 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Quetiapine fumarate
  Other Names: Seroquel

SUMMARY:
The purpose of this study is to demonstrate superior efficacy of Quetiapine fumarate sustained release (SEROQUEL) compared with placebo when used as a mono-therapy in the treatment of Major Depressive Disorders PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to provide written informed consent before beginning any study related procedures
* Patient has a documented clinical diagnosis of major depressive disorder
* Patient is able to understand and comply with the requirements of the study, as judged by a study investigator

Exclusion Criteria:

* Patients with a history of non-compliance as judged by the study investigator
* Patients with a known lack of response to previous treatment with quetiapine
* Patients who have participated in a clinical trial within 4 weeks of randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2006-04; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of Quetiapine SR compared with placebo in the treatment of patients with MDD as assessed by change from randomization to Week 8 in the MADRS total score

SECONDARY OUTCOMES:
To evaluate if Quetiapine SR improves the health-related quality of life of patients with MDD, compared to placebo
To evaluate if quetiapine SR reduces anxiety symptoms in patients with MDD, compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (34):
- United States (34):
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, El Centro, California
  - Research Site, Garden Grove, California
  - Research Site, National City, California
  - Research Site, Riverside, California
  - Research Site, Hartford, Connecticut
  - Research Site, Wilmington, Delaware
  - Research Site, Altamonte Springs, Florida
  - Research Site, DeLand, Florida
  - Research Site, Maitland, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Naperville, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Lafayette, Indiana
  - Research Site, Owensboro, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Braintree, Massachusetts
  - Research Site, Cambridge, Massachusetts
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research SIte, Staten Island, New York
  - Research Site, Avon Lake, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Allentown, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, DeSoto, Texas
  - Research Site, Houston, Texas

REFERENCES:
- [Derived] McIntyre RS, Gorwood P, Thase ME, Liss C, Desai D, Chen J, Bauer M. Early Symptom Improvement as a Predictor of Response to Extended Release Quetiapine in Major Depressive Disorder. J Clin Psychopharmacol. 2015 Dec;35(6):706-10. doi: 10.1097/JCP.0000000000000416. PMID 26474010
- [Derived] Weisler R, Montgomery SA, Earley WR, Szamosi J, Eriksson H. Extended release quetiapine fumarate in patients with major depressive disorder: suicidality data from acute and maintenance studies. J Clin Psychiatry. 2014 May;75(5):520-7. doi: 10.4088/JCP.13m08624. PMID 24816198
- [Derived] Weisler R, McIntyre RS. The role of extended-release quetiapine fumarate monotherapy in the treatment of patients with major depressive disorder. Expert Rev Neurother. 2013 Nov;13(11):1161-82. doi: 10.1586/14737175.2013.846520. PMID 24175720
- [Derived] Clayton AH, Locklear JC, Svedsater H, McIntyre RS. Sexual functioning in patients with major depressive disorder in randomized placebo-controlled studies of extended release quetiapine fumarate. CNS Spectr. 2014 Apr;19(2):182-96. doi: 10.1017/S1092852913000631. Epub 2013 Sep 25. PMID 24067192
- [Derived] Thase ME, Montgomery S, Papakostas GI, Bauer M, Trivedi MH, Svedsater H, Locklear JC, Gustafsson U, Datto C, Eriksson H. Quetiapine XR monotherapy in major depressive disorder: a pooled analysis to assess the influence of baseline severity on efficacy. Int Clin Psychopharmacol. 2013 May;28(3):113-20. doi: 10.1097/YIC.0b013e32835fb971. PMID 23485955
- [Derived] Bortnick B, El-Khalili N, Banov M, Adson D, Datto C, Raines S, Earley W, Eriksson H. Efficacy and tolerability of extended release quetiapine fumarate (quetiapine XR) monotherapy in major depressive disorder: a placebo-controlled, randomized study. J Affect Disord. 2011 Jan;128(1-2):83-94. doi: 10.1016/j.jad.2010.06.031. Epub 2010 Aug 6. PMID 20691481